CLINICAL TRIAL: NCT06610175
Title: Quantitative Imaging of Cervical Spinal Structures in Healthy Participants and Patients With Cervical Degenerative Disc Disease - the DISC Pilot Study -
Brief Title: Quantitative Imaging of Cervical Spinal Structures - the DISC Pilot Study -
Acronym: DISC
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 16948
Record Dates: First submitted 2024-05-22; First posted 2024-09-24 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cervical Radiculopathy; Cervical Myelopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy participants
  Interventions: Device: Quantitative MRI and anatomical MRI
- Patients with CDDD
  Interventions: Device: Quantitative MRI and anatomical MRI

INTERVENTIONS:
Device: Quantitative MRI and anatomical MRI — The total scanning time will be approximately 40 minutes. Additionally, 10 healthy participants and 10 patients with symptomatic CDDD will undergo a second MRI with additional sequences for assessment of reproducibility on another day/time. Also: included participants will undergo neurologic examination and fill out questionnaires for NDI, VAS-arm, VAS-neck, WA-SI, EQ-5D-5L, CSI, mJOA and Nurick.
  Other Names: zoomed-DTI, Arterial Spin Labelling (ASL), Diffusion Susceptibility Contrast (DSC), Dynamic Contrast Enhanced (DCE), Synthethic MRI (SyMRI), Tomo-MR-Elastography (TMRE)

SUMMARY:
The aim of this study is to explore a multi-parametric quantitative MRI approach to measure cervical intervertebral discs, the spinal cord and its nerve roots in healthy participants and patients with cervical degenerative disc disease (CDDD).

CDDD is the consequence of degeneration of intervertebral discs and joints leading to symptoms of cervical radiculopathy, myelopathy, or a combination of both. The incidence of symptomatic CDDD is rising with the aging population, and, consequently, a significant increase in surgeries for symptomatic CDDD is predicted in the upcoming years. However, the decision for- and optimal timing of surgery remain challenging.

Currently, the decision for surgery in patients with symptomatic CDDD is related to symptoms, as well as position and size of disc herniation on conventional Magnetic Resonance Imaging (MRI). However, conventional MRI only enables qualitative morphological evaluation, leaving space for subjective individual interpretation. Also, disc herniations on conventional MRI are frequently found in asymptomatic individuals, while, in symptomatic individuals type and extent of disc herniation does not correlate to severity of symptoms. Altogether, the current standard using conventional MRI cannot optimally predict response to surgery for patients with symptomatic CDDD.

The primary aim of this project is to investigate whether a combination of different quantitative imaging sequences can provide more detailed information on disc herniation related compression and potentially aid in determining more objective cut-offs to stage disc herniation in patients with symptomatic CDDD, as well as to analyze whether differences exist in quantitative imaging parameters of discs in healthy participants versus patients with symptomatic CDDD. These novel techniques are promising, as they are noninvasive and could potentially aid in determining objective cut-offs to stage disc herniation. Since no single measurement has been proven to be the golden standard in previous studies, it is likely that a combination of measurements is needed for clinical application

DETAILED DESCRIPTION:
RATIONALE:

Cervical degenerative disc disease (CDDD) is the consequence of degeneration of intervertebral discs and joints and can result in compression of the cervical nerve root leading to clinical symptoms of radiculopathy, compression of the spinal cord with symptoms of myelopathy, or a combination of both.The incidence of CDDD is rising with the aging population, and, consequently, a significant increase insurgeries for symptomatic CDDD is predicted in the upcoming years. As such, the decision for- and optimal timing of surgery remain challenging.

Currently, the decision for surgery in patients with symptomatic CDDD is related to symptoms, as well as position and size of disc herniation on conventional Magnetic Resonance Imaging (MRI). However, conventional MRI only enables qualitative morphological evaluation, leaving space for subjective individual interpretation. Also, disc herniations on conventional MRI are frequently found in asymptomatic individuals, while, in symptomatic individuals type and extent of disc herniation does not correlate to severity of symptoms. Altogether, the current standard using conventional MRI cannot optimally predict response to surgery for patients with symptomatic CDDD.

Quantitative imaging is rapidly being recognized as a supplement to conventional MRI and refers to the direct measurement of physical properties of tissue. These novel techniques are promising, as they are noninvasive and could potentially aid in determining objective cut-offs to stage disc herniation. Diffusion tensor imaging (DTI) is one of the most studied quantitative techniques and allows for evaluation of microstructural changes. The DTI fractional anisotropy (FA) metric was demonstrated as valid biomarker for recovery after surgery in cervical myelopathy as well as surgical selection in lumbar radiculopathy. Moreover, recent introduction of zoomed-DTI (z-DTI) could lead to greater imaging accuracy while proven feasible in the cervical spine.

Furthermore, the cervical spinal cord and its nerve roots are highly vascularized and their perfusion could be compromised by disc-herniation related compression. Using the endogenous perfusion technique arterial spin labeling (ASL), as well as contrast-based perfusion techniques such as susceptibility contrast (DSC) and dynamic contrast enhanced (DCE), degree of ischemia, hypoxia as well as signal enhancement can be estimated. ASL has been studied twice for spinal cord perfusion mapping and DSC was demonstrated feasible in the spine of healthy participants as well as patients with cervical myelopathy. Additionally, increased signal enhancement was observed for DCE in degenerative discs of the lumbar spine. To our best knowledge, no studies have been conducted to assess perfusion of the cervical nerve roots, which are compromised in cervical radiculopathy due to CDDD.

Besides microstructure and perfusion, viscoelastic properties of cervical spinal structures may change in relation to disc herniation-related compression. Therefore, it would be interesting to study mechanical properties such as stiffness and viscosity, which can be measured with Tomo-MRElastography (TMRE). To our best knowledge, no previous study has assessed cervical intervertebral discs and spinal structures using TMRE, making this a promising first study.

Finally, imaging is a relatively time-consuming matter, and including additional sequences will only increase its lengthiness. Therefore, several methods are being developed to perform imaging in a more efficient manner. One novel method is Synthetic MRI (SyMRI). Advantages of SyMRI are a reduced acquisition time, possibility of performing automatic tissue segmentation and volume estimation and acquisition of quantitative parameters. SyMRI has been studied once in the spine, and significant differences in quantitative intervertebral disc values were found in relation to hydration-status of the disc.

Since no single measurement has been proven to be the golden standard in previous studies, it is likely that a combination of measurements is needed for clinical application. Therefore, the aim of this pilot study is to explore a multi-parametric quantitative MRI approach including z-DTI, ASL, DSC, DCE, TMRE, and SyMRI to measure cervical intervertebral discs, the spinal cord and its nerve roots.

OBJECTIVE:

This study will consist of three parts. The primary objective of part 1 is to evaluate feasibility of the quantitative MRI sequences (e.g. z-DTI, ASL, DSC, DCE, TMRE, and SyMRI) for assessment of cervical spinal structures (e.g. intervertebral discs, spinal cord, and nerve roots) in healthy participants and patients with symptomatic CDDD. The primary objective of part 2 is to determine a correlation between the quantitative MRI sequences of cervical spinal structures to clinical outcome in patients with symptomatic CDDD. Finally, the primary aim of part 3 is to establish a correlation between quantitative MRI sequences of cervical spinal structures and surgical treatment within 6 months of follow-up.

STUDY DESIGN:

A prospective pilot study.

STUDY POPULATION:

The study population consists of healthy participants and patients with symptomatic CDDD with radiculopathy, myelopathy, or radiculomyelopathy. Age-matched healthy participants will be included. Participants have no previous history of cervical disc herniation or cervical surgery, a sufficient understanding of the Dutch language and no contraindications for an MRI scan.

INTERVENTION:

All participants will be subjected to several MRI sequences, using a state of the art 3T Siemens MRI Scanner available in the UMCG. First, all participants (healthy participants and patients with symptomatic CDDD) undergo baseline neurologic examination. Additionally, participants fill out the following questionnaires: Neck Disability Index (NDI), Visual Analogue Scale (VAS) for arm and neck pain, modified Japanese Orthopedic Association (mJOA), Nurick grade, EuroQol 5-Dimension 5-Level (EQ-5D-5L), Work Ability Single Item (WAI-SI), and Central Sensitisation Inventory (CSI). All participants undergo MRI scanning: localizer & T2-weighted anatomical (conventional MRI), z-DTI, ASL, DSC, DCE, TMRE, and SyMR. The total scanning time will be approximately 40 minutes. For assessment of reproducibility, 10 healthy participants and 10 patients will be scanned 2 times on different days/times. The patients with symptomatic CDDD will have another study visit after 6 months of follow-up to assess their treatment status (having had surgery yes/no; in case of yes also the surgery characteristics), to fill out the abovementioned questionnaires and have an MRI with additional sequences.

MAIN STUDY PARAMETERS/ENDPOINTS:

Primary endpoints are the technical feasibility and repeatability for the quantitative MRI sequences (i.e. z_DTI, ASL, DSC, DCE, TMRE, and SyMRI) of cervical spinal structures (i.e. intervertebral discs, spinal cord, and nerve roots) in healthy participants and patients with symptomatic CDDD. Also, a correlation of quantitative MRI sequences of cervical spinal structures to clinical impairment in patients with symptomatic CDDD will be determined. Clinical impairment will be measured with the Neck Disability Index (NDI) for cervical radiculopathy, modified Japanese Orthopaedic Association Score (mJOA) for cervical myelopathy, and NDI as well as mJOA for radiculomyelopathy.

NATURE AND EXTENT OF THE BURDER AND RISKS ASSOCIATED WITH PARTICIPATION, BENEFIT AND GROUP RELATEDNESS:

All participants (healthy and patients) will need a conventional MRI scan with quantitative MRI sequences, which will take approximately 40 minutes. Most MRI sequences used in this study are noninvasive and do not involve any ionizing radiation. However, DSC and DCE require administration of a bolus contrast. The contrast agent that will be used is Dotarem. Without any contra-indications for an MRI scan or contrast agent, health is not at risk. There is an overall negligible risk for participants, as based on the Risk Classification Checklist of the NFU. Therefore, the investigators can conclude that this study is a low-risk study.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic CDDD

* Age ≥18 years
* One-level or 2-level symptomatic CDDD (radiculopathy, myelopathy or radiculomyelopathy) of cervical levels C4-5, C5-6l, C6-7 or C7-Th1.
* Sufficient understanding of spoken and written Dutch language
* Agrees to participate in the obligatory measurements of this study and signed informed consent prior to any study-related procedures.
* Women who use anticonception or are in their menopause. If this is not the case, a negative pregnancy test is necessary.

Healthy participants

* Age-matched healthy participant.
* Sufficient understanding of spoken and written Dutch language.
* Agrees to participate in the obligatory measurements of this study and signed informed consent prior to any study-related procedures.
* Women who use anticonception or are in their menopause. If this is not the case, a negative pregnancy test is necessary

Exclusion Criteria:

Patients with symptomatic CDDD

* Multi-segmental (3 or more segments) symptomatic CDDD.
* Contraindication for an MRI scan (e.g. implanted non-MRI-compatible devices or foreign bodies, claustrophobic or pregnancy).
* A positive pregnancy test.
* Allergy for contrast medium.
* Previous history of cervical spine surgery.

Healthy participants

* Contraindication for an MRI scan (e.g. implanted non-MRI-compatible devices or foreign bodies, claustrophobic or pregnancy).
* A positive pregnancy test.
* Allergy for contrast medium.
* Previous history of cervical spine surgery.
* Complaints of symptomatic CDDD (radiating arm/neck pain, tingling fingers, loss of strength or changed sensibility in one of the upper extremities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants and patients with symptomatic CDDD with an appointment at the neurosurgical outpatient clinic will be asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Quantitative MRI sequences | MRI conducted at study visit (baseline)
  Technical feasibility and repeatibility of quantitative MRI sequences (i.e. z-DTI, ASL, DSC, DCE, SyMRI, and TMRE) of cervical spinal structures (i.e. intervertebral disc, spinal cord, and nerve roots) in healthy participants and patients with symptomatic CDDD.
Clinical correlation of quantitative MRI sequences and clinical impairment in patients with symptomatic CDDD | MRI and clinical examinations conducted at study visit (baseline)
  To determine a correlation of quantitative MRI sequences of cervical spinal structures to clinical impairment in patients with symptomatic CDDD. Clinical impairment will be measured with the Neck Disability Index (NDI) for cervical radiculopathy, modified Japanese Orthopaedic Association Score (mJOA) for cervical myelopathy, and NDI as well as mJOA for cervical radiculomyelopathy.
To determine a correlation between baseline quantitative MRI sequences of cervical spinal structures and surgical treatment after 6 months of follow-up in patients with symptomatic CDDD as well as clinical outcomes assessed at 6 months of follow-up. | 6 months
Comparison CSI | During first study visit
  To make a comparison of the CSI-score in healthy participants with bulging discs on MRI compared to patients with symptomatic CDDD.

SECONDARY OUTCOMES:
Correlation between quantitative MRI sequences of the cervical spinal cord with extent of compression on anatomical MRI (cross-sectional area spinal cord) in healthy participants and patients with symptomatic CDDD. | Comparison made at baseline and for patients with symptomatic CDDD also at 6 months follow-up
  Extent of compression on anatomical MRI is measured as a ratio between the diameter of the spinal canal and spinal cord as well as with different shape analysis and segmentations.
Between-group analyses comparing quantitative MRI sequences of cervical spinal structures of healthy participants to subgroups of patients | MRI conducted at baseline and at 6 months follow-up in the patients with symptomatic CDDD
  Patients with symptomatic CDDD as a whole group, only patients with cervical radiculopathy, only patients with cervical myelopathy
Comparison of quantitative MRI sequences of cervical spinal structures in healthy participants and patients with symptomatic CDDD to available values in literature. | Assessed during study visit
To determine a correlation of quantitative MRI sequences of cervical spinal structures to clinical outcomes | MRI conducted at baseline and at 6 months follow-up in the patients with symptomatic CDDD
  Clinical outcomes measured with Visual Analogue Scale (VAS)-arm, VAS-neck, Nurick grade, EuroQol 5- Dimension 5-Level (EQ-5D-5L), and Work Ability Single item (WA-S

CONTACTS AND LOCATIONS:
Overall Officials: Jos Kuijlen, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided